CLINICAL TRIAL: NCT06372379
Title: Development of a Multipurpose Dashboard to Monitor the Situation of Emergency Departments. An Observational Prospective Study
Brief Title: Development of a Multipurpose Dashboard to Monitor the Situation of Emergency Departments
Acronym: eCREAM-UC2
Status: Not yet recruiting | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Astir S.r.l. (Unknown); Orobix Life S.r.l. (Unknown); Fondazione Bruno Kessler (Other)
Responsible Party: Sponsor
Other Study IDs: 8780_UC2
Record Dates: First submitted 2024-04-09; First posted 2024-04-18 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Emergency Medicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adults who attended the emergency department
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
An emergency department (ED) is a healthcare service that provides the first clinical assessment and treatment to patients with various acute conditions. These departments, however, are often overwhelmed by the large volume of patients. As a consequence, ED crowding has become a global concern and has been correlated to reduced timeliness and effectiveness of care and increased patient mortality. Concerning input, 20% to 30% of patients are brought to the ED by ambulance; the remaining are self-presenting for the vast majority. Notably, non-urgent conditions characterize a high proportion of all ED visits worldwide, and almost all of these visits involve self-presenting patients. Increasing the awareness of these patients about the mandate of EDs and the real-time situation of the neighboring emergency departments has the potential to reduce the self-presentation of patients with minor, non-urgent conditions. Such patient empowerment can be achieved through a dashboard. Concerning throughput, working in the ED requires emergency physicians and nurses to treat many patients at once while maintaining situational awareness of the surroundings. This is especially true for the head of the department, but it also holds for all physicians. It can be crucial, for example, for physicians to know if there is a bottleneck in the flow of the entire patient care process, such as a particularly high average waiting time for radiology reporting or cardiologic consultation. The availability of this information allows countermeasures to be put in place to regain efficiency. All this can be achieved through dedicated dashboards automatically fed from various information system. In addition, appropriate dashboards also enable health policymakers to monitor specific epidemiological phenomena, such as the emergence of certain infectious diseases, in a timely manner.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Arrived at emergency department between 1 January 2025 and 31 December 2025

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients who arrived at participating emergency departments between January 1, 2025 and December 31, 2025
Sampling Method: Probability Sample
Enrollment: 162000 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Daschboards | September 2024 - September 2027
  Develop three different control panels for three different end-users, specifically:
  1. Dashboard for citizens
  2. Dashboard for healthcare providers
  3. Dashboard for healthcare policymakers The aim is to extract the needed information from heterogeneous sources and to feed the dashboards according to the needs of the end-users. On the whole, for citizens, the dashboard will be designed to empower them to choose the most appropriate ED to attend or to consider a different, more relevant or more efficient, health service; for healthcare providers, the dashboard will provide a clear and immediate picture of the ED situation in terms of patient flow and workflow; for healthcare policymakers, the dashboard will provide the ability to monitor specific phenomena of interest, such as ED crowding level, possible incidence of pre-specified epidemiological phenomena, availability and timeliness of primary and secondary patient transfers, ambulance offload delays, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Guido Bertolini, MD, Principal Investigator — Istituto Di Ricerche Farmacologiche Mario Negri

IPD SHARING:
Plan to Share IPD: Yes
The anonymized data derived from this study could be shared for secondary use in the context of research projects.
Supporting Information: Study Protocol